CLINICAL TRIAL: NCT05653323
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single and Multiple-dose Escalation Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of VX-993 in Healthy Adults
Brief Title: A Phase 1 Dose Escalation Study of VX-993 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX22-993-001; 2022-002413-42 (EudraCT Number)
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A: Single Ascending Dose (SAD) (Experimental): Participants will be randomized to receive a single dose of different dose levels of VX-993.
  Interventions: Drug: VX-993
- Part B: Multiple Ascending Dose (MAD) (Experimental): Participants will be randomized to receive multiple doses of different dose levels of VX-993. The dose levels will be determined based on the data from Part A.
  Interventions: Drug: VX-993
- Placebo Part A (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-993.
  Interventions: Drug: Placebo
- Placebo Part B (Placebo Comparator): Participants will be randomized to receive multiple doses of placebo matched to VX-993.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-993 — Suspension for oral administration.
  Arms: Part A: Single Ascending Dose (SAD); Part B: Multiple Ascending Dose (MAD)
Drug: Placebo — Suspension for oral administration.
  Arms: Placebo Part A; Placebo Part B

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of VX-993 at different doses in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight of more than (>) 50 kg
* Participants of non-childbearing potential
* Nonsmoker or ex-smoker for at least 3 months before screening

Key Exclusion Criteria:

* History of febrile illness or other acute illness within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 25
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 25
Part B: Safety and Tolerability as Assessed by Number of Participants With Clinically Meaningful Findings in Columbia Suicide Severity Rating Scale (C-SSRS) Responses | Pre-dose up to Day 25

SECONDARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of VX-993 | Pre-dose up to Day 25
Part B: Maximum Observed Plasma Concentration (Cmax) of VX-993 | Pre-dose up to Day 25
Part A: Area Under the Concentration Versus Time Curve (AUC) of VX-993 | Pre-dose up to Day 25
Part B: Area Under the Concentration Versus Time Curve (AUC) of VX-993 | Pre-dose up to Day 25
Part B: Pain Tolerance Threshold (PTT) for the Cold Pressor Test | Day 1, Day 10, and Day 11

CONTACTS AND LOCATIONS:
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing